CLINICAL TRIAL: NCT07242573
Title: Evaluation of the Effect of Individualized Physical Training and Neuromodulation on Pain, Sleep and Fatigue in Patients With Fibromyalgia: a Randomized Controlled Trial
Brief Title: Effect of Physical Exercise and Neuromodulation on Pain, Sleep and Fatigue in Patients With Fibromyalgia: a Randomized Controlled Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIGRR
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome (CFS)
Keywords: Fibromyalgia; Rehabilitation; Sleep Quality; Pain Management; Exercise Therapy; NESA X-Signal; Transcutaneous Electrical Stimulation; Neuromodulation; Physiotherapy; Physical Training; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Sleep Initiation and Maintenance Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to three parallel groups:
  1. Physical training using the Zebris treadmill and Alfa balance platform,
  2. Transcutaneous neuromodulation with the NESA X-Signal device,
  3. Control group with conventional physiotherapy only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Physical Training Group (Experimental): Participants receive a structured physical training program using the Zebris diagnostic treadmill and Alfa balance platform, combined with conventional physiotherapy. Sessions are conducted 5 times per week for 3 weeks and include aerobic, balance, and coordination exercises tailored individually to each patient.
  Interventions: Other: Physical Training Program
- 2. Neuromodulation Group (Experimental): Participants undergo non-invasive transcutaneous neuromodulation (NESA X-Signal) combined with conventional physiotherapy. Sessions last 30 minutes and are performed 5 times per week for 3 weeks.
  Interventions: Device: NESA X-Signal
- 3. Control Group (Active Comparator): Participants receive conventional physiotherapy only, including general exercise therapy, manual therapy, laser therapy, and relaxation sessions, consistent with standard clinical care for fibromyalgia patients.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Physical Training Program — Structured physical training using Zebris diagnostic treadmill and Alfa balance platform, performed under physiotherapist supervision. Sessions are held 5 times per week for 3 weeks and include aerobic, balance, and coordination exercises tailored to individual patient needs.
  Arms: 1. Physical Training Group
Device: NESA X-Signal — Non-invasive transcutaneous neuromodulation using the NESA X-Signal device. The device delivers microcurrent stimulation through gloves and socks electrodes (25 total) to modulate autonomic nervous system activity and reduce pain. Sessions last 30 minutes, performed 3 times per week for 6 weeks.
  Arms: 2. Neuromodulation Group
Other: Conventional Physiotherapy — Standard physiotherapy program consisting of general exercise therapy, relaxation and breathing training, manual therapy, and light physical modalities (e.g., laser, heat therapy). No neuromodulation or device-based interventions are applied.
  Arms: 3. Control Group

SUMMARY:
Fibromyalgia (FMS) is a chronic, multifactorial syndrome characterized by widespread pain, fatigue, and cognitive disturbances. This interventional study evaluates the impact of structured physical training using diagnostic-training devices (Zebris treadmill and Alfa balance platform) and transcutaneous neuromodulation (NESA X-Signal) on pain, sleep quality, and overall health status in patients with fibromyalgia and chronic fatigue symptom.

Participants are allocated into three groups:

1. Physical training + conventional physiotherapy,
2. Transcutaneous neuromodulation + conventional physiotherapy,
3. Control (conventional physiotherapy only). The results will support the development of evidence-based rehabilitation protocols for fibromyalgia patients.

DETAILED DESCRIPTION:
The study is conducted at the National Institute of Geriatrics, Rheumatology, and Rehabilitation (NIGRiR), Warsaw, Poland. It includes 75 patients aged 20-80 years with a confirmed diagnosis of fibromyalgia and chronic fatigue symptom. Participants are randomly assigned to one of three groups:

Group 1 receives structured physical training using the Zebris treadmill and Alfa balance platform, along with conventional physiotherapy.

Group 2 undergoes non-invasive transcutaneous neuromodulation (NESA X-Signal) and conventional physiotherapy.

Group 3 serves as a control group, receiving conventional physiotherapy only.

The interventions last 6 weeks, supervised by a multidisciplinary rehabilitation team. Clinical evaluations include pain intensity (VAS, WPI, SSS), fatigue (FSS, FIS), sleep quality (PSQI), depressive symptoms (Beck Depression Scale), and functional mobility assessments.

Data are analyzed statistically to compare within- and between-group differences. The study aims to determine the effectiveness of combined exercise and neuromodulation programs in improving physical and psychological well-being among fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years
* Confirmed diagnosis of fibromyalgia
* Presence of chronic fatigue symptoms
* Stable health condition
* Presence of sleep disturbances
* Ability to provide written informed consent and cooperate during the study

Exclusion Criteria:

* Lack of informed consent or cooperation
* Refusal to undergo procedures beyond standard NFZ physiotherapy
* Cancer
* Neurological disorders (e.g., neuralgia, multiple sclerosis, diabetic polyneuropathy, stroke)
* Diagnosed dementia or cognitive impairment
* Implanted electronic devices (e.g., pacemaker)
* Internal bleeding or acute febrile illness
* Acute thrombophlebitis
* Hysteria or electric phobia
* Neurotic addiction to stimulation
* Infectious skin diseases (e.g., mycosis, purulent dermatitis)
* Inability to communicate in Polish sufficiently to complete questionnaires or follow instructions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity (Visual Analogue Scale - VAS 0-10) | Baseline to 6 weeks (post-intervention)
  Difference in VAS pain score between baseline and post-intervention across study arms.
Change in sleep quality (Pittsburgh Sleep Quality Index - PSQI) | Baseline to 6 weeks (post-intervention)
  Change in PSQI global score from baseline to post-intervention across study arms.

SECONDARY OUTCOMES:
Change in depressive symptoms (Beck Depression Inventory - BDI) | Baseline to 6 weeks
  Change in BDI total score from baseline to post-intervention.
Change in Widespread Pain Index (WPI) and Symptom Severity Scale (SSS) | Baseline to 6 weeks
  Change in ACR diagnostic components (WPI and SSS) between baseline and post-intervention.
Change in fatigue severity (Fatigue Severity Scale - FSS) | Baseline to 6 weeks
  Change in FSS total score from baseline to post-intervention.
Change in fatigue impact (Fatigue Impact Scale - FIS) | Baseline to 6 weeks
  Change in FIS total score assessing functional impact of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Beata Tarnacka, Professor, MD, PhD, Study Director — Rehabilitation Clinic, National Institute of Geriatrics, Rheumatology and Rehabilitation (NIGRiR), Warsaw, Poland; Justyna Frasuńska, MD, PhD, Study Chair — Rehabilitation Clinic, National Institute of Geriatrics, Rheumatology and Rehabilitation (NIGRiR), Warsaw, Poland; Filip Królikowski, MSc, Physiotherapist, Principal Investigator — Rehabilitation Clinic, National Institute of Geriatrics, Rheumatology and Rehabilitation (NIGRiR), Warsaw, Poland
Locations (1):
- Rehabilitation Clinic, National Institute of Geriatrics, Rheumatology and Rehabilitation (NIGRiR), Warsaw, Masovian Voivodeship, Poland